CLINICAL TRIAL: NCT00807482
Title: Diagnostic and Clinical Characterization of Patients With Unusual Genetic Disorders of the Airways
Brief Title: Pathogenesis of Primary Ciliary Dyskinesia (PCD) Lung Disease
Status: Recruiting | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 98-1015; 5R01HL071798 (NIH)
Record Dates: First submitted 2008-12-11; First posted 2008-12-12 (Estimated); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Kartagener Syndrome
Keywords: Primary Ciliary Dyskinesia; Mucociliary Clearance; Genetic Mutation
MeSH Terms: conditions — Kartagener Syndrome; Ciliary Motility Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, buckle scrape, semen, and scrape biopsy of nasal cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: People who have been definitively diagnosed with primary ciliary dyskinesia (PCD).

SUMMARY:
The overall short-term goals of this project include the following: 1) identify the genes that are key to the function of respiratory cilia to protect the normal lung; and 2) the effects of genetic mutations that adversely affect ciliary function and cause primary ciliary dyskinesia (PCD), which results in life-shortening lung disease. The long-term goal of this project is to develop better understanding of the underlying genetic variability that adversely modifies ciliary function, and predisposes to common airway diseases, such as asthma and chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
A key component of lung defense is the efficiency of mucociliary clearance (MCC).

Primary ciliary dyskinesia (PCD) is a human genetic disorder with defective MCC. This ongoing project is designed to identify additional disease-causing mutations in PCD, and correlate the molecular etiologies with the ciliary phenotype (ultrastructure, wave form and beat frequency). We have recently shown that the normal human cilium has a distinctive waveform, i.e. beats in-plane with defined curvatures and amplitudes for the effective (forward) and recovery stroke. We hypothesize that discrete sets of genes contribute to the structure and function of the ciliary outer dynein arm (ODA), inner dynein arm (IDA), and central pair (CP) and radial spoke (RS) complex (CP/RS), and that we can identify novel genetic mutations in different structural components of the cilium that will have different effects on ciliary ultrastructure, wave form, and beat frequency. Importantly, we are now able to identify patients with PCD who do not have hallmark diagnostic ultrastructural defects, based on distinctive clinical phenotypes (including situs inversus), low or borderline nasal NO production, and abnormal ciliary motility. Identification of PCD patients with normal ciliary ultrastructure (~16% of PCD patients at UNC) offers the opportunity to discover mutations in genes that cause functional, but not ultrastructural, defects (such as DNAH11), and to correlate those mutations with ciliary waveform abnormalities. Over the past 4 years, we have made great progress in identifying mutations in 2 genes (DNAI1 and DNAH5) that cause ~60% of ODA defects in PCD, and ~35% of PCD overall. We will extend our search for disease causing mutations in PCD, using several different approaches, including studies of additional candidate genes, (guided by ultrastructure), plus insights from ciliary proteomics, and family-based studies. Taken together, these studies will provide new insights regarding the relationship of mutations in specific genes to ciliary ultrastructural and functional defects. These studies will not only greatly enhance our ability to diagnose PCD, but will also lead to discovery of "milder" genetic mutations associated with normal ciliary ultrastructure, and likely some residual ciliary function. Ultimately, this will allow future studies of the role of partial loss of ciliary function in the predisposition to more common airways diseases, such as chronic bronchitis and chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a high suspicion for the diagnosis of PCD, based on clinical features

Healthy Volunteers who have a family member with confirmed PCD.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have a high suspicion for the diagnosis of PCD, based on clinical features.
Sampling Method: Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2004-01; Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
This is not an interventional study | This is not an interventional study
  Not applicable. This is not an interventional study.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth R. Olivier, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Noone PG, Zariwala MB,Knowles MR. Primary Ciliary Dyskinesia. In: Principles of Molecular Medicine. Editors: MS Runge and C Patterson, 2nd Edition, Humana Press, Totowa, NJ, pp 239-250, 2006.
- [Background] Knowles MR, Leigh MW, Ostrowski LE, Huang L, Carson JL, Hazucha MJ, Yin W, Berg JS, Davis SD, Dell SD, Ferkol TW, Rosenfeld M, Sagel SD, Milla CE, Olivier KN, Turner EH, Lewis AP, Bamshad MJ, Nickerson DA, Shendure J, Zariwala MA; Genetic Disorders of Mucociliary Clearance Consortium. Exome sequencing identifies mutations in CCDC114 as a cause of primary ciliary dyskinesia. Am J Hum Genet. 2013 Jan 10;92(1):99-106. doi: 10.1016/j.ajhg.2012.11.003. Epub 2012 Dec 20. PMID 23261302
- [Result] Zariwala MA, Leigh MW, Ceppa F, Kennedy MP, Noone PG, Carson JL, Hazucha MJ, Lori A, Horvath J, Olbrich H, Loges NT, Bridoux AM, Pennarun G, Duriez B, Escudier E, Mitchison HM, Chodhari R, Chung EM, Morgan LC, de Iongh RU, Rutland J, Pradal U, Omran H, Amselem S, Knowles MR. Mutations of DNAI1 in primary ciliary dyskinesia: evidence of founder effect in a common mutation. Am J Respir Crit Care Med. 2006 Oct 15;174(8):858-66. doi: 10.1164/rccm.200603-370OC. Epub 2006 Jul 20. PMID 16858015
- [Result] Hornef N, Olbrich H, Horvath J, Zariwala MA, Fliegauf M, Loges NT, Wildhaber J, Noone PG, Kennedy M, Antonarakis SE, Blouin JL, Bartoloni L, Nusslein T, Ahrens P, Griese M, Kuhl H, Sudbrak R, Knowles MR, Reinhardt R, Omran H. DNAH5 mutations are a common cause of primary ciliary dyskinesia with outer dynein arm defects. Am J Respir Crit Care Med. 2006 Jul 15;174(2):120-6. doi: 10.1164/rccm.200601-084OC. Epub 2006 Apr 20. PMID 16627867
- [Result] Kennedy MP, Noone PG, Leigh MW, Zariwala MA, Minnix SL, Knowles MR, Molina PL. High-resolution CT of patients with primary ciliary dyskinesia. AJR Am J Roentgenol. 2007 May;188(5):1232-8. doi: 10.2214/AJR.06.0965. PMID 17449765
- [Result] Kennedy MP, Omran H, Leigh MW, Dell S, Morgan L, Molina PL, Robinson BV, Minnix SL, Olbrich H, Severin T, Ahrens P, Lange L, Morillas HN, Noone PG, Zariwala MA, Knowles MR. Congenital heart disease and other heterotaxic defects in a large cohort of patients with primary ciliary dyskinesia. Circulation. 2007 Jun 5;115(22):2814-21. doi: 10.1161/CIRCULATIONAHA.106.649038. Epub 2007 May 21. PMID 17515466
- [Result] Zariwala MA, Knowles MR, Omran H. Genetic defects in ciliary structure and function. Annu Rev Physiol. 2007;69:423-50. doi: 10.1146/annurev.physiol.69.040705.141301. PMID 17059358
- [Result] Lie H, Zariwala MA, Helms C, Bowcock AM, Carson JL, Brown DE 3rd, Hazucha MJ, Forsen J, Molter D, Knowles MR, Leigh MW, Ferkol TW. Primary ciliary dyskinesia in Amish communities. J Pediatr. 2010 Jun;156(6):1023-1025. doi: 10.1016/j.jpeds.2010.01.054. Epub 2010 Mar 29. PMID 20350728
- [Result] Berg JS, Evans JP, Leigh MW, Omran H, Bizon C, Mane K, Knowles MR, Weck KE, Zariwala MA. Next generation massively parallel sequencing of targeted exomes to identify genetic mutations in primary ciliary dyskinesia: implications for application to clinical testing. Genet Med. 2011 Mar;13(3):218-29. doi: 10.1097/GIM.0b013e318203cff2. PMID 21270641
- [Result] Ferkol TW, Puffenberger EG, Lie H, Helms C, Strauss KA, Bowcock A, Carson JL, Hazucha M, Morton DH, Patel AC, Leigh MW, Knowles MR, Zariwala MA. Primary ciliary dyskinesia-causing mutations in Amish and Mennonite communities. J Pediatr. 2013 Aug;163(2):383-7. doi: 10.1016/j.jpeds.2013.01.061. Epub 2013 Mar 7. PMID 23477994
- [Result] Daniels ML, Leigh MW, Davis SD, Armstrong MC, Carson JL, Hazucha M, Dell SD, Eriksson M, Collins FS, Knowles MR, Zariwala MA. Founder mutation in RSPH4A identified in patients of Hispanic descent with primary ciliary dyskinesia. Hum Mutat. 2013 Oct;34(10):1352-6. doi: 10.1002/humu.22371. Epub 2013 Aug 6. PMID 23798057
- [Result] Zariwala MA, Gee HY, Kurkowiak M, Al-Mutairi DA, Leigh MW, Hurd TW, Hjeij R, Dell SD, Chaki M, Dougherty GW, Adan M, Spear PC, Esteve-Rudd J, Loges NT, Rosenfeld M, Diaz KA, Olbrich H, Wolf WE, Sheridan E, Batten TF, Halbritter J, Porath JD, Kohl S, Lovric S, Hwang DY, Pittman JE, Burns KA, Ferkol TW, Sagel SD, Olivier KN, Morgan LC, Werner C, Raidt J, Pennekamp P, Sun Z, Zhou W, Airik R, Natarajan S, Allen SJ, Amirav I, Wieczorek D, Landwehr K, Nielsen K, Schwerk N, Sertic J, Kohler G, Washburn J, Levy S, Fan S, Koerner-Rettberg C, Amselem S, Williams DS, Mitchell BJ, Drummond IA, Otto EA, Omran H, Knowles MR, Hildebrandt F. ZMYND10 is mutated in primary ciliary dyskinesia and interacts with LRRC6. Am J Hum Genet. 2013 Aug 8;93(2):336-45. doi: 10.1016/j.ajhg.2013.06.007. Epub 2013 Jul 25. PMID 23891469
- [Result] Tarkar A, Loges NT, Slagle CE, Francis R, Dougherty GW, Tamayo JV, Shook B, Cantino M, Schwartz D, Jahnke C, Olbrich H, Werner C, Raidt J, Pennekamp P, Abouhamed M, Hjeij R, Kohler G, Griese M, Li Y, Lemke K, Klena N, Liu X, Gabriel G, Tobita K, Jaspers M, Morgan LC, Shapiro AJ, Letteboer SJ, Mans DA, Carson JL, Leigh MW, Wolf WE, Chen S, Lucas JS, Onoufriadis A, Plagnol V, Schmidts M, Boldt K; UK10K; Roepman R, Zariwala MA, Lo CW, Mitchison HM, Knowles MR, Burdine RD, Loturco JJ, Omran H. DYX1C1 is required for axonemal dynein assembly and ciliary motility. Nat Genet. 2013 Sep;45(9):995-1003. doi: 10.1038/ng.2707. Epub 2013 Jul 21. PMID 23872636
- [Result] Hjeij R, Lindstrand A, Francis R, Zariwala MA, Liu X, Li Y, Damerla R, Dougherty GW, Abouhamed M, Olbrich H, Loges NT, Pennekamp P, Davis EE, Carvalho CM, Pehlivan D, Werner C, Raidt J, Kohler G, Haffner K, Reyes-Mugica M, Lupski JR, Leigh MW, Rosenfeld M, Morgan LC, Knowles MR, Lo CW, Katsanis N, Omran H. ARMC4 mutations cause primary ciliary dyskinesia with randomization of left/right body asymmetry. Am J Hum Genet. 2013 Aug 8;93(2):357-67. doi: 10.1016/j.ajhg.2013.06.009. Epub 2013 Jul 11. PMID 23849778
- [Result] Funkhouser WK 3rd, Niethammer M, Carson JL, Burns KA, Knowles MR, Leigh MW, Zariwala MA, Funkhouser WK Jr. A new tool improves diagnostic test performance for transmission em evaluation of axonemal dynein arms. Ultrastruct Pathol. 2014 Aug;38(4):248-55. doi: 10.3109/01913123.2013.815081. Epub 2013 Aug 19. PMID 23957500
- [Result] Knowles MR, Ostrowski LE, Loges NT, Hurd T, Leigh MW, Huang L, Wolf WE, Carson JL, Hazucha MJ, Yin W, Davis SD, Dell SD, Ferkol TW, Sagel SD, Olivier KN, Jahnke C, Olbrich H, Werner C, Raidt J, Wallmeier J, Pennekamp P, Dougherty GW, Hjeij R, Gee HY, Otto EA, Halbritter J, Chaki M, Diaz KA, Braun DA, Porath JD, Schueler M, Baktai G, Griese M, Turner EH, Lewis AP, Bamshad MJ, Nickerson DA, Hildebrandt F, Shendure J, Omran H, Zariwala MA. Mutations in SPAG1 cause primary ciliary dyskinesia associated with defective outer and inner dynein arms. Am J Hum Genet. 2013 Oct 3;93(4):711-20. doi: 10.1016/j.ajhg.2013.07.025. Epub 2013 Sep 19. PMID 24055112
- [Result] Leigh MW, Hazucha MJ, Chawla KK, Baker BR, Shapiro AJ, Brown DE, Lavange LM, Horton BJ, Qaqish B, Carson JL, Davis SD, Dell SD, Ferkol TW, Atkinson JJ, Olivier KN, Sagel SD, Rosenfeld M, Milla C, Lee HS, Krischer J, Zariwala MA, Knowles MR. Standardizing nasal nitric oxide measurement as a test for primary ciliary dyskinesia. Ann Am Thorac Soc. 2013 Dec;10(6):574-81. doi: 10.1513/AnnalsATS.201305-110OC. PMID 24024753
- [Result] Austin-Tse C, Halbritter J, Zariwala MA, Gilberti RM, Gee HY, Hellman N, Pathak N, Liu Y, Panizzi JR, Patel-King RS, Tritschler D, Bower R, O'Toole E, Porath JD, Hurd TW, Chaki M, Diaz KA, Kohl S, Lovric S, Hwang DY, Braun DA, Schueler M, Airik R, Otto EA, Leigh MW, Noone PG, Carson JL, Davis SD, Pittman JE, Ferkol TW, Atkinson JJ, Olivier KN, Sagel SD, Dell SD, Rosenfeld M, Milla CE, Loges NT, Omran H, Porter ME, King SM, Knowles MR, Drummond IA, Hildebrandt F. Zebrafish Ciliopathy Screen Plus Human Mutational Analysis Identifies C21orf59 and CCDC65 Defects as Causing Primary Ciliary Dyskinesia. Am J Hum Genet. 2013 Oct 3;93(4):672-86. doi: 10.1016/j.ajhg.2013.08.015. PMID 24094744